CLINICAL TRIAL: NCT04868981
Title: To Evaluate the Tolerability, Pharmacodynamics and Pharmacokinetics of GST-HG141 Tablets in Multiple-center, Randomized, Double-blind, Placebo-controlled Multiple-dose, Multiple-administration Study in Patients With Chronic Hepatitis B
Brief Title: Study on the Tolerability, Pharmacodynamics and Pharmacokinetics of GST-HG141 Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fujian Cosunter Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GST-HG141-21-01
Record Dates: First submitted 2021-04-23; First posted 2021-05-03 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2021-04

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GST-HG141 (Experimental): GST-HG141 tablets at varying dosages by mouth for 28 days
  Interventions: Drug: GST-HG141 tablets
- Matching Placebo for GST-HG141 (Placebo Comparator): Placebos for GST-HG141 tablets at varying dosages by mouth for 28 days
  Interventions: Drug: Matching Placebos for GST-HG141 tablets

INTERVENTIONS:
Drug: GST-HG141 tablets — Administrate GST-HG141 tablets orally in fed state twice daily at 25 mg or 50mg or 100 mg doses
  Arms: GST-HG141
Drug: Matching Placebos for GST-HG141 tablets — Administrate the placebos for GST-HG141 tablets orally in fed state twice daily at 25 mg or 50mg or 100 mg doses
  Arms: Matching Placebo for GST-HG141

SUMMARY:
To Evaluate the Tolerability, Pharmacodynamics and Pharmacokinetics of GST-HG141 Tablets in Multiple-center, Randomized, Double-blind, Placebo-controlled Multiple-dose, Multiple-administration Study in Patients With Chronic Hepatitis B (CHB)

DETAILED DESCRIPTION:
This study includes 3 cohorts of 25 mg BID, 50 mg BID and 100 mg BID. 30 patients with chronic hepatitis B will be enrolled in this study and each cohort will enroll 10 patients (GST-HG141 tablets : PBO=8:2). All enrolled patients will be given research drugs twice a day for 28 days (D28 was administered only once in the morning). And each cohort requires at least 4 subjects with elevated ALT. Tolerability, pharmacodynamics and pharmacokinetics will be evaluated according to the protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent before the study and fully understand the content and process of the study as well as the possible adverse drug reactions;
2. Be able to complete the study in accordance with protocol requirements;
3. Subjects (including partners) are willing to take effective contraceptive measures from completion of screening to 6 months after the last Administration;
4. Ages ranged from 18 to 70 years old (including 18 and 70 years old);
5. Male subjects weighing no less than 45 kg, and female subjects weighing no less than 40 kg. [Body mass index (BMI) = body weight (kg) / height 2 (m^2)], body mass index is in the range of 18 ~ 32 kg / m^2 (including critical value);
6. Patients with HBsAg-positive for at least 6 months (based on outpatient/inpatient medical records or laboratory report; or with IgM HBcAb-negative and HBsAg-positive when screening;
7. Patients without interferon/nucleoside analogue treatment when screening, or interferon treatment was stopped more than 1 year ago, and nucleoside analogue treatment was stopped more than 6 months ago.
8. For HBeAg-positive patients, HBV DNA ≥ 2×10^5 IU/mL; For HBeAg-negative patients, HBV DNA ≥ 2×10^4 IU/mL;
9. Patients with Serum ALT less than 5×ULN when screening.

Exclusion Criteria:

1. Patients with suspected allergy to any component of the study drug or allergic constitution (multiple drug and food allergy)；
2. Patients who had major trauma or Large surgical operation within 3 months before screening or are planning to take surgical treatment during the study ;
3. Patients who had blood donation or massive blood loss (≥400 mL), or had a blood transfusion within 3 months before screening; or had blood donation or massive blood loss (≥200 mL) within 1 months before screening;
4. Patients with smoking more than 5 cigarettes per day within 3 months before the study or heavy drinking within 4 weeks before screening (drinking more than 14 units of alcohol per week: 1 unit = 285 mL of beer, or 25 mL of spirits, or 100 mL of wine)；
5. Patients who had used immunosuppressants, immunomodulators (thymosin) and cytotoxic drugs within 6 months before dosing, or had received live attenuated vaccine within 1 month before screening;
6. Patients who used immunosuppressants, immunomodulators (thymosin) and cytotoxic drugs within 6 months before dosing, or who had received live attenuated vaccine within 1 month before screening;
7. Patients with clinically significant acute or chronic liver disease caused by non HBV infection (fatty liver disease is ruled out or recruited by researcher);
8. Patients with history of liver cirrhosis or progressive liver fibrosis (e.g., liver histopathology reported liver cirrhosis or endoscopy indicated esophageal and gastric varices);
9. Patients with confirmed or suspected decompensated hepatitis B cirrhosis including but not limited to: hepatic encephalopathy, hepatorenal syndrome, esophageal and gastric variceal bleeding, splenomegaly, ascites, primary liver cancer, etc. ;
10. Patients with history of other malignancies or complicating with other malignant tumors;
11. Patients complicating with severe circulatory, digestive, respiratory, urinary, blood, metabolism, immune, nervous and other systemic;
12. Patients with acute infection within 2 weeks before screening;
13. Patients who had participated in clinical trials of drugs or medical devices within 1 month before screening;
14. Patients who could not ban smoking, drinking, caffeinated food or drinks within 2 days before administration and during the study , and patients who have special dietary requirements and can not follow the unified diet;
15. Laboratory examination: platelet count<90×10^9/L; leukocyte count<3.0×10^9/L; neutrophil absolute value<1.3×10^9/L; serum total bilirubin>2×ULN; albumin<30 g/L; creatinine clearance rate≤60ml/min (calculated by MDRD formula); international standardization ratio value of prothrombin time (INR) >1.5;
16. Patients with Alpha fetoprotein (AFP) more than 50 UG / L or imaging findings of malignant liver lesions;
17. Patients with HCAb-positive , AIDS Ag/Ab-positive, or positive syphilis spirochemical Ab simultaneously RPR test-positive;
18. For patients with normal ALT or less than 2×ULN, LSM≥12.4 kPa; or for patients with ALT≥2×ULN, LSM≥17.0 kPa;
19. Patients with positive urine drug screening (morphine, marijuana) or alcohol breath test;
20. Patients with positive urine drug screening (morphine, marijuana) or alcohol breath test；
21. Patients with other factors that are not suitable to participate in this study in researcher's thought.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-05-31 (Actual); Primary Completion 2022-02-23 (Actual); Study Completion 2022-03-14 (Actual)

PRIMARY OUTCOMES:
Number of patients with chronic HBV infection with treatment-related adverse events and laboratory abnormalities. | Up to 33 days
  Symptoms and physical examination, clinical laboratory examination, vital signs，12 lead ECG and adrenal ultrasounds were collected and assessed by CTCAE v5.0.
Cmax of GST-HG141 | Measured on -0.5, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12hours on Day1; -0.5 hours on Day 8, Day 15, Day22 and Day 27 for trough concentration; -0.5, 0.5 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours on Day 28.
  Plasma samples were collected at different points for pharmacokinetic analysis
AUC of GST-HG141 | Measured on -0.5, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12hours on Day1; -0.5 hours on Day 8, Day 15, Day22 and Day 27 for trough concentration; -0.5, 0.5 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours on Day 28.
  Plasma samples were collected at different points for pharmacokinetic analysis
t1/2 of GST-HG141 | Measured on -0.5, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12hours on Day1; -0.5 hours on Day 8, Day 15, Day22 and Day 27 for trough concentration; -0.5, 0.5 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours on Day 28.
  Plasma samples were collected at different points for pharmacokinetic analysis
Cl/F of GST-HG141 | Measured on -0.5, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12hours on Day1; -0.5 hours on Day 8, Day 15, Day22 and Day 27 for trough concentration; -0.5, 0.5 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours on Day 28.
  Plasma samples were collected at different points for pharmacokinetic analysis

SECONDARY OUTCOMES:
The value of serum HBV DNA decreased from baseline | Plasma samples were collected before administation on the morning of day 1 and day 15 and at any time on day 29 and day 33
  Plasma samples were collected at different points for pharmacodynamics analysis
The value of serum HBV pgRNA decreased from baseline | Plasma samples were collected before administation on the morning of day 1 and day 15 and at any time on day 29 and day 33
  Plasma samples were collected at different points for pharmacodynamics analysis
The value of serum HBsAg decreased from baseline | Plasma samples were collected before administation on the morning of day 1 and day 15 and at any time on day 29 and day 33
  Plasma samples were collected at different points for pharmacodynamics analysis
The value of serum HBeAg decreased from baseline | Plasma samples were collected before administation on the morning of day 1 and day 15 and at any time on day 29 and day 33
  Plasma samples were collected at different points for pharmacodynamics analysis

CONTACTS AND LOCATIONS:
Overall Officials: Junqi Niu, PhD, Principal Investigator — The First Hospital of Jilin University
Locations (1):
- The first hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wu M, Mai J, Zhang H, Zhang G, Mao J, Tang Y, Yan W, Wu W, Hou J, Liang X, Liu Z, Ding Y, Niu J. Safety, pharmacokinetics, and antiviral efficacy of the novel capsid assembly modulator GST-HG141 in patients with chronic hepatitis B: a phase 1 trial with a randomized, placebo-controlled design. Virol J. 2024 Dec 20;21(1):328. doi: 10.1186/s12985-024-02584-8. PMID 39707469